CLINICAL TRIAL: NCT00720161
Title: Metformin in Children With Motor Deficit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ML3830
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2011-09

CONDITIONS: Spina Bifida; Neuromuscular Diseases
Keywords: metformin, spina bifida, duchenne, insulin resistance
MeSH Terms: conditions — Spinal Dysraphism; Neuromuscular Diseases; Muscular Dystrophy, Duchenne; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Metformin during 12 months and then 6 months Placebo (Active Comparator): Metformin during 12 months and then 6 months Placebo
  Interventions: Drug: Metformin; Drug: Placebo
- B: Placebo during 6 months, afterwards 12 months metformin (Placebo Comparator): Placebo during 6 months, afterwards 12 months metformin
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Metformin — daily 850 mg
Drug: Placebo — placebo

SUMMARY:
Obesity with insulin resistance in the paediatric population provides an increasing challenge. Children with neurological or neuromuscular diseases are even more prone to obesity: their locomotor impairment leads to an increasingly sedentary lifestyle, a decrease in physical fitness and an increase in body fat (1-3). Obesity, in turn, can be associated with a decrease in physical fitness and a further increase in body fat. In this study we want to evaluate the effect of an insulin-sensitizer, metformin, in a group of overweight/obese patients with neurological or neuromuscular diseases. Metformin is a well-established insulin sensitizer.

DETAILED DESCRIPTION:
Obesity with insulin resistance in the paediatric population provides an increasing challenge. Children with neurological or neuromuscular diseases are even more prone to obesity: their locomotor impairment leads to an increasingly sedentary lifestyle, a decrease in physical fitness and an increase in body fat (1-3). Obesity, in turn, can be associated with a decrease in physical fitness and a further increase in body fat. In this study we want to evaluate the effect of an insulin-sensitizer, metformin, in a group of overweight/obese patients with neurological or neuromuscular diseases. Metformin is a well-established insulin sensitizer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurogenic or myogenic motor deficit, clinically obese or who had excessively gained weight over the last year.

Exclusion Criteria:

* Exclusion criteria were known type 1 or type 2 diabetes mellitus and contraindications to metformin therapy.

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2006-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 12 months
  changes in insulin, fasting glucose and insulin resistance after 6 months Metformine versus 6 months placebo

SECONDARY OUTCOMES:
fat | 12 months
  changes in cholesterol and triglycerides after 6 months Metformine versus 6 months placebo

CONTACTS AND LOCATIONS:
Overall Officials: kristina m casteels, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Brabant, Belgium

REFERENCES:
- [Background] Srinivasan S, Ambler GR, Baur LA, Garnett SP, Tepsa M, Yap F, Ward GM, Cowell CT. Randomized, controlled trial of metformin for obesity and insulin resistance in children and adolescents: improvement in body composition and fasting insulin. J Clin Endocrinol Metab. 2006 Jun;91(6):2074-80. doi: 10.1210/jc.2006-0241. Epub 2006 Apr 4. PMID 16595599